CLINICAL TRIAL: NCT06954974
Title: THE EFFECT OF SMARTPHONE APPLICATION HOME-BASED EXERCISES ON SLEEP QUALITY, FATIGUE, FUNCTIONAL CAPACITY, AND QUALITY OF LIFE IN OBSTRUCTIVE SLEEP APNEA IN JEDDAH
Brief Title: SMARTPHONE APPLICATION HOME-BASED EXERCISES IN OBSTRUCTIVE SLEEP APNEA IN JEDDAH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Mohanad Ayfan, MOHANAD AYFAN, Coordinator Physical Therapy Track. Faculty of Medical Rehabilitation Sciences, KAU, KSA., King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: physical therapy and osa
Record Dates: First submitted 2025-01-29; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: OSA - Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Exercise Therapy; Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- exercise alone (Experimental)
  Interventions: Other: Exercise
- CPAP device and exercise. (Experimental)
  Interventions: Device: CPAP device and exercise
- CPAP device alone (Experimental)
  Interventions: Device: CPAP device

INTERVENTIONS:
Device: CPAP device — CPAP device
  Arms: CPAP device alone
Device: CPAP device and exercise — CPAP device
  Arms: CPAP device and exercise.
Other: Exercise — 1. Retropalatal level: Phase I: • Open your mouth • Pronounce "A" for 5 seconds • Stop. Close your mouth. Procedure: 2 sets of 10 repetitions.
  2. Retroglossal level: Phase I: • Push the tongue against the front of the palate • Move it back to perform a "click" sound, Phase II: • Move the tongue from right to left and from up to down The sequence of movement directions can be randomized to increase the challenge for repetitions., Phase III: • In this exercise, the tongue of the patient will scroll • Circle with the tongue on the inside of the lips • Draw 10 circles per set.
     Phase IV: • pressing the back of the tongue firmly on the oral cavity's floor for 8 seconds. Phase V: • Step 1, bite the tongue depressor. • Step 2, push the tongue against the tongue depressor and hold for 8 seconds. Procedure: 2 sets of 10 repetitions.
  3. Deglutition level: Phase I: • Gently hold the tongue between the front teeth • Maintain this position Then, close your mouth and swallow. Phase II: • This vers
  Arms: exercise alone

SUMMARY:
The study aim is to explore the effects of a home-based exercise training smartphone application on sleep quality, fatigue, functional capacity, and quality of life among obstructive sleep apnea (OSA) patients in Jeddah city, Saudi Arabia.

DETAILED DESCRIPTION:
"Obstructive sleep apnea" (OSA) explains upper airway blockage episodes that recur frequently as you sleep and cause sporadic hypoxia, daytime sleepiness, and impaired cognitive performance. If treatment is not received, OSA can have severe effects on the cardiovascular system and can be fatal . Obesity is one of the significant risk factors for OSA, and it is twice as common in obese individuals as in those of typical weight . Additionally, it has been shown that obesity and the apnea-hypopnea index (AHI) are correlated; a 10% rise in weight is linked to a 32% increase in the AHI . Although the Always the first treatment for Although People who have OSA require constant positive airway pressure, there is mounting evidence that weight loss can also mitigate the severity of OSA .

In Saudi Arabia, Between December 2005 and March 2006, surveys were undertaken by the University of King Khalid and the King Fahd National Guard Primary Health Clinics in Riyadh to ascertain The rate of OSA symptoms in the People of middle age. The study found that OSA symptoms were quite prevalent. One in three middle-aged Male Saudis are susceptible to OSA in the primary care setting .

The upper airway repeatedly collapsing or constricting while you sleep is the primary reason behind both apnea and hypopnea in patients with OSA. Therefore, limiting upper airway collapse may theoretically help to alleviate the problem of apnea/hypopnea during sleep. Recent research indicates that both morphological and non-anatomical variables may be involved in the upper airway collapse when you sleep . OSA can have a significant detrimental effect on life quality (QoL) and is linked to several health issues, such as daytime tiredness, exhaustion, fatigue, depression, functional and cognitive decline that can increase the duration of sedentary time, and cardiovascular diseases .

Polysomnography is the gold standard for diagnosing OSA (PSG).The majority popular and extensively used tool to assess the intensity of OSA is the apnea and hypopnea index (AHI), which PSG offers. The total of all episodes (hypopneas and apneas) divided by the number of sleep hours is the AHI. Values between 5 and 14 are classified as mild, those between 15 and 29 as a medium, and those higher Thirty as severe.

Oral-pharyngeal rehabilitation can reduce Sleep apnea and its severity in some cases by maintaining the upper airway open and improving the tensile strength, rigidity and reactivity of the neck, tongue, and muscles governing the soft palate's mobility, both intrinsic and extrinsic..These findings are supported by case-control research that showed persons with poor sleep quality had lower levels of physical activity than comparable adults without sleep issues. For example, compared to people without sleep apnea, persons with OSA had a lower likelihood of being active, and longitudinal and cross-sectional data indicate that those who exercise frequently have a lower prevalence and incidence of OSA . The fatigue and sleepiness, as well as the extra weight and poor energy characteristic of the clinical presentation of OSA and the accompanying neurocognitive changes, have been linked to the low levels of physical activity reported in these individuals.

For many rehabilitation programs, the at-home exercise regimen is crucial. . This is especially true in light of the COVID-19 epidemic, as many regions may view hospital visits for rehabilitation as superfluous. The Natural home rehabilitation, however, requires that the person completes physical therapy activities on their own, unsupervised by a licensed physical therapist or other medical experts. As a result, the patient's recollection or the helping family member or caregiver frequently account for all of the performance quality, which is not the best course of action for any physical activity program. In the therapeutic community, smartphone applications for at-home rehabilitation programs have gained a lot of attention. Numerous research have looked into how smartphone apps affect older persons' activity, fall prevention, and Parkinsonism. .

However, to our knowledge, there isn't a program, gadget, or application made to help people with OSA carry out at-home rehabilitation exercises. The OSA rehabilitation program necessitates a certain amount of ability in contrast to programs that primarily target gross motor abilities, such as those for fall prevention or Parkinson's disease. .

The aim of the present thesis is to explore the effects of a home-based exercise training smartphone application on sleep quality, fatigue, functional capacity, and quality of life among obstructive sleep apnea (OSA) patients in Jeddah city, Saudi Arabia.

In the present thesis, the investigators hypothesize that using a home-based exercise training smartphone application will improve OSA patients' outcomes, including sleep quality, fatigue, functional capacity, and quality of life among OSA patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with confirmed mild or moderate OSA
* aged between 18 and 65 years
* BMI ≤ 40 kg/m2
* agreed to participatein the study were recruited.

Exclusion Criteria:

* Pregnant patients
* individuals younger than 18 or older than 65
* those who refused to participate in the study
* those with severe cardiopulmonary conditions such as chronic obstructive pulmonary disease or heart failure
* those with head and neck anomalies
* those with a BMI >40 kg/m² were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-25 (Estimated); Primary Completion 2025-11-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Assessment | BASE LINE - 3 MONTH
  The Short Form 36 (SF-36) questionnaire was used to measure the Health-Related Quality of Life (HRQOL) at baseline and at follow-up. The SF-36 was selected because of its capacity to assess quality of life in both physical and psychological domains. It is considered a standard instrument for evaluating HRQOL and was created by Ware and Sherbourne in the United States.
  The 36 items on the questionnaire are broken down into eight domains. The ability to carry out daily tasks including walking, taking care of oneself, and relaxing is assessed by the Physical Functioning (PF) domain, which comprises items 3 through 11. The role restrictions due to physical problems (RP) domain, which includes items 12 through 15, looks at how role constraints and everyday activities are impacted by physical issues. Items 20 to 21 make up the Bodily Pain (BP) domain, which gauges how much pain has interfered with everyday activities and how severe it has been throughout the previ
Sleep Quality | BASE LINE - 3 MONTH
  The Pittsburgh Sleep Quality Index (PSQI), created by Buysse et al., was used to evaluate the quality of sleep in each group. The PSQI is a self-reported instrument that assesses seven aspects of sleep quality over a month: subjective sleep quality, sleep latency, length, habitual sleep efficiency, sleep disruptions, use of sleep aids, and dysfunction during the day. The majority of the 19 items on the PSQI are answered on a Likert scale. Component scores, which range from 0 to 3, are produced by combining these items. A score of "0" indicates no sleep issues at all and score of "3" denotes serious sleep issues.
  For instance, the daytime dysfunction score is calculated from two items: the frequency of medication use for sleep and the frequency of trouble staying awake during daily activities such as driving or eating. These items are coded on a scale of 0 to 3 (0 = no issues, 1-2 = mild issues, 3-4 = moderate issues, 5-6 = severe issues). The subjective sleep quali
Fatigue | BASE LINE - 3 MONTH
  The Fatigue Severity Scale (FSS) was used to measure the patient's level of fatigue.. Each of the nine FSS items, which rate the degree of fatigue symptoms and their impact on patient functioning (such as motivation, exercise, physical functioning, carrying out duties, and interfering with work, family, or social life), is given a score between 1 (completely disagree) and 7 (completely agree). The questions include statements like "my fatigue is very debilitating" and "exercise brings on my fatigue." For every item, a higher score denotes a higher level of fatigue. All patients who responded to at least half of the FSS items had their scores determined using the conventional scoring procedure for the FSS, which involves averaging the nine items to provide an overall score that ranges from 1 (no fatigue) to 7 (very severe fatigue). A FSS average score of < 4 is considered non fatigue, while a score ≥ 4 indicates fatigue.
Functional Capacity | BASE LINE - 3 MONTH
  The 6-minute walk test (6MWT) is a widely utilized tool for assessing functional exercise capacity, particularly in patients with moderate to severe cardiovascular conditions. This test was employed in this study to measure the patients' functional capacity. The 6MWT is a straightforward and practical test that only requires a 100-foot hallway, with no specialized exercise equipment or advanced training for the administering technicians. Since walking is a common activity for nearly all patients, except those with severe impairments, the test measures the maximum distance a patient can walk in six minutes on a flat, hard surface. It evaluates the combined responses of various systems involved in exercise, including the pulmonary, cardiovascular, and peripheral circulatory systems, blood, neuromuscular units, and muscle metabolism. Unlike maximal cardiopulmonary exercise testing, the 6MWT does not provide detailed insights into the function of individual organs or
Sleep Test Results | BASE LINE - 3 MONTH
  (AHI): The total number of apnea and hypopnea episodes that transpire throughout each hour of sleep is known as the AHI. A considerable decrease in breathing lasting at least 10 seconds is known as a hypopnea, while a total stop or cessation of breathing lasting at least 10 seconds is known as an apnoea. When combined, apnea and hypopnea cause mini-awakenings and oxygen level dips that interfere with sleep. The frequency of apnea and hypopnea per hour is a measure of the severity of sleep apnea. It is classified as normal (0-5 events/hour), mild (5-15 events/hour), moderate (15-30 events/hour), and severe (> 30 events/hour) by the American Academy of Sleep Medicine (AASM).
  Sleep Efficiency: The percentage of time spent sleeping compared to the amount of time spent in bed is known as sleep efficiency. The percentage is computed by dividing the total amount of time spent in bed by the total amount of sleep. A sleep efficiency of 80% or above is regarded as normal.
BMI | BASE LINE - 3 MONTH
  (weight and height will be combined to report BMI in kg/m^2). weight in kilograms, height in meters